CLINICAL TRIAL: NCT00855777
Title: Evaluation of Analgesic Efficacy of Etoricoxib Compared With Ibuprofen in Third Molar Extraction Pain.
Brief Title: Etoricoxib Versus Ibuprofen in Third Molar Extraction Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: professor Roberto Corrocher, Department of Clinical and Experimental Medicine - University of Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Verona - CE1597
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-03

CONDITIONS: Dental Extraction
Keywords: third molar extraction; etoricoxib; ibuprofen; analgesic efficacy; pain
MeSH Terms: conditions — Pain | interventions — Etoricoxib; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etoricoxib (Experimental): Etoricoxib 120 mg/day x 3 days
  Interventions: Drug: etoricoxib
- Ibuprofen (Active Comparator): Ibuprofen 1800 mg/day x 3 days
  Interventions: Drug: ibuprofen

INTERVENTIONS:
Drug: etoricoxib — etoricoxib 120 mg/day for 3 days
  Arms: Etoricoxib
Drug: ibuprofen — ibuprofen 1,800 mg/day for 3 days
  Arms: Ibuprofen

SUMMARY:
The aim of this study is to evaluate the analgesic efficacy of etoricoxib compared with a well known and widely used non-steroid antinflammatory drug, ibuprofen, in third molar extraction pain. At this time, there are no data about the efficacy of etoricoxib for reducing pain following dental extraction.

This will be a single center, randomized, double-blind study, in which patients with moderate to severe pain following third molar extraction will be randomized to receive etoricoxib (120 mg in a single dose + 2 dose of placebo pro day for 3 days) or ibuprofen (1800 mg in 3 doses pro day for 3 days). Paracetamol plus codeine will be used as rescue medication. Pain assessment will be performed using a 11-point pain intensity scale (0 = no pain and 10 = worster pain) during the first 3 days after dental extraction. Patients will be enrolled 15 days before the dental extraction. During enrollment visit a complete clinical evaluation with particular attention for potential exclusion criteria (e.g. hypertension and cardiovascular risk factors) as well as blood analyses will be performed. A follow-up visit will be performed 15 days after the dental extraction. Tolerability will be assessed through recording of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* subjects with age > 18 years
* in good health status (assessed in occasion of enrollment visit) without any major systemic illness
* candidate to third molar extraction and presenting local pain within 2 hours after dental extraction

Exclusion Criteria:

* patients with any major systemic illness
* patients with a clinical history of drug abuse
* patients with hypertension and/or a condition of increased cardiovascular risk
* pregnant or lactating women
* patients with a history of hypersensitivity/allergy to analgesic drugs, including classical NSAID or coxibs
* patients with either high levels of liver enzymes (major of 1.5x the upper limit of reference interval) or of creatinine(major of 1.2x the upper limit of reference interval)
* patients with either a history of peptic ulcer or of haemorrhagic diathesis
* patients who can not ensure an adequate compliance for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
analgesic efficacy | 3 days

SECONDARY OUTCOMES:
side effects | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Corrocher, MD, Study Director — Universita di Verona